CLINICAL TRIAL: NCT02567877
Title: Is Levothyroxine Alone Adequate Thyroid Hormone Replacement for All Patients?
Brief Title: Is Levothyroxine Alone Adequate Thyroid Hormone Replacement?
Status: Terminated | Type: Observational
Why Stopped: poor enrollment
Sponsor: University of Colorado, Denver (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Other Study IDs: 14-2155; UL1TR001082 (NIH)
Record Dates: First submitted 2015-10-01; First posted 2015-10-05 (Estimated); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Postsurgical Hypothyroidism; Hypothyroidism
Keywords: hypothyroidism; deiodinase polymorphism; cognitive function; thyroidectomy; levothyroxine
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroidectomy; Thyroxine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- levothyroxine in thyroidectomy patients: patients undergoing thyroidectomy for nodular thyroid disease
  Interventions: Procedure: thyroidectomy; Drug: levothyroxine in thyroidectomy patients

INTERVENTIONS:
Procedure: thyroidectomy — Patients enrolled in the study will undergo a clinically-indicated thyroidectomy performed as standard of care.
  Other Names: near-total thyroidectomy; total thyroidectomy
Drug: levothyroxine in thyroidectomy patients — Patients will initiate levothyroxine treatment after surgery consistent with standard of care. The drug dosage will be titrated to TSH goal that matches the pre-surgery TSH (+/- 1 mIU/L)
  Other Names: Synthroid; Levothyroid; Tirosint

SUMMARY:
Patients taking thyroid hormone replacement after thyroid removal surgery often report feeling differently than they did prior to taking thyroid hormone. The symptoms can include fatigue, worsening mood or subjective "brain fog" where the patient feels like their thinking is just not as sharp as it was previously. Multiple studies have found that patients taking thyroid hormone replacement have a diminished quality of life compared to matched controls. Previous studies have suggested that the type of deiodinase (DIO) polymorphism a patient has, which is responsible for converting the thyroid hormone T4 into the more biologically active T3, may contribute to their overall cognition and sense of well-being. The Investigators aim to determine if the type of deiodinase polymorphism a patient has contributes to the patient's cognition and overall sense of well-being after surgery and thyroid hormone replacement.

Objective: Determine if patients with the deiodinase type 2 CC polymorphism have objective differences in working memory (N-back test is primary endpoint), cognitive function and sense of well-being after thyroidectomy when placed on standard thyroid hormone replacement therapy.

Hypotheses: (1) Patients with the deiodinase type 2 CC polymorphism will have worse working memory (N-back test is primary endpoint), cognitive function and sense of well-being on standard thyroid hormone replacement therapy after thyroidectomy compared with before thyroidectomy.

(2) Patients with the deiodinase type 2 TT or TC polymorphism will have no differences in working memory, cognitive function or sense of well-being on standard thyroid hormone replacement before and after thyroidectomy.

DETAILED DESCRIPTION:
STUDY DESIGN Many patients undergo thyroidectomy for nodular thyroid disease. They have normal thyroid function prior to surgery and are immediately placed on standard thyroid hormone replacement therapy (levothyroxine, LT4) after surgery. The levothyroxine dose is titrated every 6-8 weeks to normalize the thyroid stimulating hormone (TSH) level. The investigators aim to study this population before surgery when the patients still have endogenous thyroid function and after surgery once their TSH has been normalized to pre-surgery levels. Using a weight based dosing strategy (1.6mcg/kg), most patients will remain euthyroid throughout this process. This experimental design eliminates many of the confounding variables that have plagued previous thyroid replacement trials. One of the most difficult aspects of conducting these types of studies is testing a uniform patient population. The most common cause of hypothyroidism is autoimmune thyroiditis (Hashimoto's thyroiditis) and previous studies have largely focused on these patients. The difficulty in testing patients with autoimmune thyroid failure is that even though they have a common illness, the disease course is extremely variable. Each patient may have different degrees of thyroid failure and may still be making different amounts of endogenous thyroid hormone. The presence of thyroid autoantibodies has also been reported to have systemic effects, and may influence perception of overall health and sense of well-being. This study will focus on a more homogenous population without the potential cofounders inherent to patients with autoimmune thyroid disease. Each patient will serve as their own control and also avoid any cognitive or somatic effects that temporary hypothyroidism may induce.

No study has ever evaluated a patient's symptoms before and after replacement with thyroid hormone when the patient is euthyroid before thyroid hormone therapy. The assumption has been made that if serum TSH is normalized, thyroid hormone levels are adequate and that symptoms of hypothyroidism have been relieved. The investigators know from large community based studies that symptoms of hypothyroidism persist despite what the investigators believe is "adequate" thyroid hormone replacement in as many as 10% of patients. Our study will be the first to test the same patient, before and after thyroidectomy so the investigators can directly compare normal endogenous thyroid function with levothyroxine (LT4) therapy resulting in the same serum TSH. Thyroidectomies are often performed for large nodules or nodules that show indeterminate or suspicious cytology after fine needle aspiration biopsy, but turn out to be benign at final histological diagnosis. The current standard of care is to replace thyroid hormone with LT4 to normalize the serum TSH. Our approach uses the same patient as their own control and eliminates numerous variables that cannot be controlled for in other studies including: variable onset of hypothyroidism, degree of endogenous thyroid function and underlying cause of hypothyroidism.

Prior to and after surgery, the investigators will measure each patient's thyroid levels (TSH, free T4, total T4, total T3, thyroxine binding globulin, sex hormone binding globulin, lipid panel, and iron), and parathyroid/calcium function (parathyroid hormone, calcium, albumin, vitamin D25), and deiodinase type 2 polymorphism status will be determined on pre-surgery bloodwork. Thyronamine levels will also be measured before and after surgery. Thyronamines are thyronergic metabolites of thyroid hormones that can decrease metabolism and induce behavioral inactivity in mouse models. A recently developed sensitive chemiluminescent antibody assay for 3-Iodothyronamine has been developed and patients on levothyroxine therapy after thyroidectomy had higher thyronamine levels compared with euthyroid controls. Based on these studies, the investigators hypothesize, as a secondary measure that patients with a higher thyronamine level after surgery, or greater pre- vs post-surgery thyronamine level will have worse outcomes, defined by the questionnaires. Patients will complete a series of questionnaires (SF-36 measure of overall health, Billewicz measure of thyroid health, HADS measure of anxiety and depression) as well as undergo working memory testing using the N-back and cognitive function testing using the Sustained Attention to Response Test (SART). Lab analysis will also be performed before surgery to look at targets of thyroid hormone action including low density lipoprotein (LDL) cholesterol and sex hormone binding globulin (SHBG). Following surgery, only patients benign results or low-risk differentiated thyroid cancer not requiring radioiodine therapy or TSH suppression will continue on the study. The patients continuing in the study will have their dose of levothyroxine titrated with the goal of matching their pre-surgery TSH +/- 1 milli-international units per liter (mIU/L). 6 months following surgery, lab testing, questionnaires and cognitive testing will be repeated. Timing the second set of testing 6 months will allow adequate time to match the post-surgery TSH to the pre-surgery level and give adequate time for any cognitive effects resulting from the surgery itself to dissipate. The primary endpoint will compare changes in scores on the N-back test before and after surgery from those in the deiodinase CC polymorphism group to those in the deiodinase type 2 TC and TT groups. Secondary endpoints will include scores on the SART and well-being questionnaires before and after surgery to correlate with deiodinase polymorphisms as well as correlation of these outcome measures with serum thyronamine levels before and after surgery as an exploratory measure.

An optional sub-study is being made available to research subjects to compare the stool microbiota longitudinally, with the initial stool sample at the start of the study in the presence of normal systemic thyroid hormone levels and then again after thyroidectomy while taking oral levothyroxine. Comparisons of any microbiota compositional changes from before and after surgery will be made to any changes in symptoms, cognition/memory testing and overall quality of life. Any exposure to antibiotics, probiotics or other updates to medical history will be documented at each visit. Any exposure to systemic antibiotics in the previous 60 days of the first study collection or between collections will be excluded. Subjects will complete a 3-day lead-in dietary log prior to each stool collection, summarizing meal compositions on 3 consecutive days before the stool sample is collected and submitted. Participants will be given their own dietary log again and encouraged to follow a similar diet prior to the second stool collection.

ELIGIBILITY:
Inclusion Criteria:

* TSH in the ideal reference range (0.4-4.0 milli-international units per liter (mIU/L))
* Planned thyroidectomy for nodular thyroid disease or low-risk differentiated thyroid cancer (<4cm, no ETE, no expected use of RAI or suppressive levothyroxine therapy)

Exclusion Criteria:

* History of psychiatric illness (major illness as defined by DSM IV: major depression, schizophrenia, mania, etc). Patients prescribed chronic medications for psychiatric illness, those taking benzodiazepines or anti-seizure medication.
* Estrogen therapy that is new within the last 6 weeks or if the dose has been changed within the last 6 weeks
* Positive thyroid antibodies
* Chronic use (>4 weeks) of concomitant medications that could affect cognition and memory (including sedative hypnotics, selective serotonin reuptake inhibitors, selective serotonin-norepinephrine reuptake inhibitors, Topamax, benzodiazepines, etc.)
* Pregnancy
* Steroid therapy
* Persistent cancer of any type or other major medical illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing thyroidectomy for nodular thyroid disease or low-risk thyroid cancer
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Change in working memory (N-back testing) and correlation with deiodinase type 2 polymorphism | 6-8 months
  Change in working memory as assessed by pre- vs post-surgery N-back test scores will be measured and compared between those with the deiodinase type 2 CC polymorphism versus those in the deiodinase type 2 TC and TT polymorphism group

SECONDARY OUTCOMES:
Change in cognitive function (SART testing) and correlation with deiodinase type 2 polymorphism | 6-8 months
  Changes in cognitive function assessed by SART testing pre- and post-surgery will be compared between those with the deiodinase type 2 CC polymorphism versus those in the deiodinase type 2 TC and TT polymorphism group
Change in Well-being (SF-36, Billewicz, HADS testing) and correlation with deiodinase type 2 polymorphism | 6-8 months
  Changes in well-being will be assessed with the SF-36, Billewicz, and HADS tests pre- and post-surgery will be compared between those with the deiodinase type 2 CC polymorphism versus those in the deiodinase type 2 TC and TT polymorphism group
Correlation of working memory (N-back testing) and correlation with serum thyronamine levels | 6-8 months
  Pre- vs post-surgery N-back test scores will be measured and correlated with pre- and post-surgery serum thyronamine levels
Change in cognitive function (SART testing) and correlation with serum thyronamine levels | 6-8 months
  Cognitive function assessed by SART testing pre- and post-surgery will be determined and correlated with pre- and post-surgery serum thyronamine levels
Change in Well-being (SF-36, Billewicz, HADS testing) and correlation with serum thyronamine levels | 6-8 months
  Well-being will be assessed with the SF-36, Billewicz, and HADS tests pre- and post-surgery and will be correlated with serum thyronamine levels pre- and post-surgery
Change in serum thyronamine levels | 6-8 months
  changes in serum thyronamine levels from pre-surgery to end of study (post-surgery) will be assessed
Change in sex hormone binding globulin (SHBG) | 6-8 months
  changes in serum sex hormone binding globulin levels from pre-surgery to end of study (post-surgery) will be assessed
Change in LDL cholesterol | 6-8 months
  changes in serum LDL levels from pre-surgery to end of study (post-surgery) will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Bryan R Haugen, M.D., Principal Investigator — University of Colorado Denver Anschutz Medical Campus
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

REFERENCES:
- [Background] Saravanan P, Chau WF, Roberts N, Vedhara K, Greenwood R, Dayan CM. Psychological well-being in patients on 'adequate' doses of l-thyroxine: results of a large, controlled community-based questionnaire study. Clin Endocrinol (Oxf). 2002 Nov;57(5):577-85. doi: 10.1046/j.1365-2265.2002.01654.x. PMID 12390330
- [Background] Scanlan TS, Suchland KL, Hart ME, Chiellini G, Huang Y, Kruzich PJ, Frascarelli S, Crossley DA, Bunzow JR, Ronca-Testoni S, Lin ET, Hatton D, Zucchi R, Grandy DK. 3-Iodothyronamine is an endogenous and rapid-acting derivative of thyroid hormone. Nat Med. 2004 Jun;10(6):638-42. doi: 10.1038/nm1051. Epub 2004 May 16. PMID 15146179
- [Background] Hoefig CS, Kohrle J, Brabant G, Dixit K, Yap B, Strasburger CJ, Wu Z. Evidence for extrathyroidal formation of 3-iodothyronamine in humans as provided by a novel monoclonal antibody-based chemiluminescent serum immunoassay. J Clin Endocrinol Metab. 2011 Jun;96(6):1864-72. doi: 10.1210/jc.2010-2680. Epub 2011 Apr 13. PMID 21490071
- [Background] Samuels MH, Schuff KG, Carlson NE, Carello P, Janowsky JS. Health status, mood, and cognition in experimentally induced subclinical hypothyroidism. J Clin Endocrinol Metab. 2007 Jul;92(7):2545-51. doi: 10.1210/jc.2007-0011. Epub 2007 May 1. PMID 17473069